CLINICAL TRIAL: NCT05530759
Title: Integrated Genomics and Patient-Derived Cancer Models
Brief Title: Examining Blood and Tissue Samples to Identify Diagnostic Markers in Patients With Metastatic Cancer Undergoing Tumor Removal
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 21-008623; NCI-2022-03313 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2022-08-31; First posted 2022-09-07 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Hematopoietic and Lymphoid System Neoplasm; Metastatic Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood, tissue and buccal samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (biospecimen collection): Patients undergo collection of blood and buccal samples before or after SOC biopsy or tumor resection. Patients undergo collection of tumor tissue at time of SOC biopsy or tumor resection. Patients' medical records are also reviewed. Patients' archived tissue or blood samples may also be collected.
  Interventions: Procedure: Biopsy Specimen; Procedure: Biospecimen Collection; Other: Medical Chart Review

INTERVENTIONS:
Procedure: Biopsy Specimen — Undergo collection of tissue samples
  Other Names: Biopsy Sample
Procedure: Biospecimen Collection — Undergo collection of blood and buccal swab samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Biospecimen Collection — Undergo collection of archived tissue and blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Medical Chart Review — Review of medical record
  Other Names: Chart Review

SUMMARY:
This study characterizes deoxyribonucleic acid (DNA) and proteomic (protein) changes in both biopsies and tumors removed during surgery of patients who have been diagnosed with aggressive/metastatic (that has spread to other places in the body) cancer in order to identify possible diagnostic markers and potential drugs for treating aggressive tumor types. Proteomic analyses include looking at the proteome, or all the proteins expressed, or made by DNA at a specific moment in time. Studying samples of blood, buccal (cheek), and tissue in the laboratory from patients undergoing surgical resection or biopsy may help doctors learn more about the changes that occur in the proteome, DNA alterations, and identify molecular biomarkers for which therapeutic drugs may exist. Studying the DNA in tumor tissue and in blood may also help researchers see if the tumor has important differences.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To understand the pathogenesis, molecular mechanisms, and disease processes of malignancies.

II. To examine the utility of integrated genomics for discovery of targets or pathways involved in tumor/malignancy progression of patients with malignancies.

III. To observe for any evidence of anti-tumor activity from treatment if selected based on integrated genomics.

IV. To create and offer opportunities for targeted individualized therapy based on the outcome of integrated genomics and micro-cancer modeling.

V. To determine the outcome of patients with malignancies who received targeted individualized therapy.

OUTLINE: This is an ancillary-correlative study.

Patients undergo collection of blood and buccal samples before or after standard of care (SOC) biopsy or tumor resection. Patients undergo collection of tumor tissue at time of SOC biopsy or tumor resection. Patients' medical records are also reviewed. Patients' archived tissue or blood samples may also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients (or the legally authorized representative/guardian signing on behalf of the participant) must understand and provide written informed consent prior to initiation of any study-specific procedures
* >= 18 years of age
* Patients must have a diagnosis of confirmed malignancy
* Patient is a good medical candidate for a standard of care biopsy or surgical procedure to obtain tissue or has archival tissue available for analysis

Exclusion Criteria:

* Uncontrolled concurrent illness including psychiatric illness, or situations that would limit compliance with the study requirements or the ability to willingly give written informed consent
* Inaccessible tumor for biopsy or patient does not have tumor tissue available for research use
* Biopsy must not be considered to be more than minimal risk to the patient. Contraindications to percutaneous biopsy:

  * Significant coagulopathy that cannot be adequately corrected
  * Severely compromised cardiopulmonary function or hemodynamic instability
  * Lack of a safe pathway to the lesion
  * Inability of the patient to cooperate with, or to be positioned for, the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be identified internally through provider referrals most commonly from providers in Medical Oncology.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-06-29 (Actual); Primary Completion 2027-04-07 (Estimated); Study Completion 2028-04-07 (Estimated)

PRIMARY OUTCOMES:
Deoxyribonucleic acid (DNA) alterations | Through study completion; up to five years
  identify molecular targets for which therapeutic drugs may exist
Proteomic changes in both biopsies and resected tumors | Through study completion; up to five years
  identify molecular targets for which therapeutic drugs may exist

CONTACTS AND LOCATIONS:
Overall Officials: Aaron S. Mansfield, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials